CLINICAL TRIAL: NCT07087106
Title: Novel Assessment of Glucose Consumption in Multiple Sclerosis Utilizing [F-18]FDG-PET
Brief Title: Glucose Consumption in MS Using [F-18]FDG-PET
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, TARUN SINGHAL, Associate Professor of Neurology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025P000883
Record Dates: First submitted 2025-06-13; First posted 2025-07-25 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; FDG; Positron Emission Tomography; PET
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PMS, RRMS, and Healthy Control subjects (Experimental)
  Interventions: Drug: [F-18]FDG

INTERVENTIONS:
Drug: [F-18]FDG — PET radiopharmaceutical

SUMMARY:
Given the need for better diagnostic imaging techniques in multiple sclerosis (MS), the study aims to investigate the utility of [F-18]FDG positron emission tomography (PET) in MS. The study will be assessing glucose consumption patterns in subjects with progressive MS (PMS) and relapsing-remitting MS (RRMS), as well as healthy controls. PET will be compared to magnetic resonance imaging (MRI) lesion load and brain atrophy, and serum and blood biomarkers, as well as clinical measures of physical disability, cognitive impairment, fatigue, and depression. This study's findings may pave a path for integrating [F-18]FDG-PET in routine clinical practice for MS, improving patient experiences and outcomes.

The specific aims of the study are:

Aim 1: To compare glucose consumption in the brain in subjects with PMS, relapsing-remitting MS (RRMS), and healthy controls, using the radiolabeled glucose analogue 18-fluorodeoxyglucose, also known as [F-18]FDG.

Aim 2: To compare the relationship between FDG-PET and standard 3T MRI measures including global and regional brain atrophy and lesion load, and to compare FDG-PET with MRI in terms of their relationship with clinical measures of physical disability, cognitive impairment, fatigue and depression in MS subjects.

Aim 3: To assess the relationship of FDG-PET with serum and blood biomarkers, including but not limited to sNfL, GFAP, IL-6, and TNFα in MS.

DETAILED DESCRIPTION:
This is a single center, cross-sectional study of the measurement of glucose consumption using [F-18]FDG-PET in subjects with progressive MS as compared to RRMS and healthy controls.

Three groups of subjects will be recruited:

1. Subjects meeting the definition for PMS, (secondary progressive MS (SPMS) or primary progressive MS (PPMS), by International Panel Criteria
2. Subjects meeting the definition for RRMS by the International Panel Criteria,
3. Healthy Controls

Sample Size: The investigators plan to enroll 50 subjects including 20 with PMS (SPMS or PPMS), 20 with RRMS and 10 healthy controls.

In order to attain the goal sample size of 50 subjects, the investigators estimate that they may need to consent approximately 60 subjects to account for screen failures.

Physicians at the Brigham MS Center may present the study to a subject during a regular scheduled clinic visit. If the subject is interested in the study, a copy of the consent form will be given. The subject will then be contacted by telephone prior to the screening visit appointment. At the time of the subject's screening visit, an investigator will go over the study in detail, answer any questions the subject may have regarding the study and a licensed physician investigator will obtain informed consent. Subjects will also be recruited through the MGB Rally website (https://rally.massgeneralbrigham.org). In accordance with NIH guidelines, efforts will be made to attain a mix of study participants, in terms of gender and racial/ethnic representation.

Subjects may be required to come for up to 3-4 visits for this study.

Initial Visit:

During the first visit, subjects will be administered the screening questionnaire (if that has not already been done over telephone). Subjects will review and eventually sign the consent form. They will be administered standardized questionnaires for cognitive testing and/or other co-morbidities.

Blood samples will be drawn and stored for future immunophenotyping and/or other blood assays in the future including but not limited to sNfL and GFAP.

PET Visit:

All subjects will undergo one visit for the PET scan. During the PET scan visits, all women subjects of child bearing age will undergo a stat quantitative serum hCG pregnancy test (or urine pregnancy test) and only women with a negative test will undergo the radiopharmaceutical injection.

PET imaging procedures

For PET scanning, an intravenous (IV) catheter will be inserted into the radial antecubital or other arm or hand vein for injection of tracer. Radiopharmaceutical will be injected as a bolus (up to approximately 10mCi for [F-18]FDG followed by 5 mL of saline).

The whole PET session will last up to 60-120 mins.

MRI Visit:

All subjects will undergo a 3T Brain MRI during an MRI visit that may precede or follow the PET scan visit.

Pregnancy screening prior to MRI:

All women will be queried about their pregnancy status, use of contraception and last menstrual period. If they are reliably using contraception, can state the timing of their last menstrual period, and do not believe they could be pregnant, the investigators will proceed with the MRI scan without pregnancy testing. If they cannot do this, then they will undergo a urine pregnancy test. If a woman is seeking pregnancy and not using contraception, she will undergo a urine pregnancy test.

MRI imaging procedures MRI scanning session will be performed at Brigham and Women's Hospital (BWH) MRI facility at 60 Fenwood Road, Boston, MA, using the same high-resolution acquisition protocol.

Several pulse sequences will be performed to image the brain. There will be no intravenous contrast used for the MRIs.

The MRI scan session will take up to approximately 45-60 mins.

There will be a follow up phone call within 24-72 hours after the PET scans to ensure the subjects have not suffered from any side effects.

A non-diagnostic computed tomography (CT) scan or MR scan will be performed for attenuation correction of PET transmission data at the time of initiation of scanning.

For the PET portion, as this drug is radioactive, the subject will be exposed to a small amount of radiation as a result of participation in this study. The per unit radiation dose for [F-18]FDG is 0.019 mSv/mCi (0.514 μSv/MBq). The total amount of radiation exposure from [F-18]FDG is 8mSv (for 10mCi injected dose). This amount of radiation is approximately 16% of the yearly amount of radiation allowed for persons who work with radiation. Additional dose from low dose CT performed for attenuation correction of PET images is estimated to be up to 1mSv per CT scan. Hence, the total radiation exposure from the procedure is up to 9mSv or approximately 18% of the yearly amount of radiation exposure allowed for persons working with radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years.
2. Subjects meeting the definition for MS (including SPMS, RRMS or PPMS) by International Panel (2017 McDonald) Criteria. Age and sex-matched healthy controls will also be recruited.
3. Subjects willing to undergo PET and MRI imaging.
4. Subjects willing and able to give informed consent.

Exclusion Criteria:

1. Individuals with a known alternate neurologic disorder, previous head injury, or substance abuse.
2. Individuals with a known alternate neuropsychiatric disorder, including bipolar disease and schizophrenia.
3. Concurrent medical conditions that contraindicate study procedures
4. Women who are pregnant or nursing. Also, any woman who is seeking to become pregnant or suspects she is pregnant will be excluded from enrollment.
5. Claustrophobia
6. Non-MRI compatible implanted devices.
7. Corticosteroid treatment in the past four weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PET measurements in individuals with PMS, RRMS, and healthy controls | Baseline
  To compare PET measurements including standardized uptake value (SUV) and standardized uptake value ratio (SUVR) in individuals with PMS, RRMS, and healthy controls.

SECONDARY OUTCOMES:
Correlations between PET measurements and clinical, MRI, and blood and serum measures | Baseline
  To examine correlations between PET measurements and clinical measures (e.g., Expanded Disability Status Scale, Timed 25 Foot Walk, Symbol Digit Modality Test), MRI measures (e.g., global atrophy, regional atrophy, lesion load), and blood and serum biomarkers (e.g., sNfL, GFAP).

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Singhal, MD, MBBS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No